CLINICAL TRIAL: NCT05231226
Title: Timing of Complete Revascularization in Patients With ST-segment Elevation Myocardial Infarction And Multivessel Disease-A Multi-center Randomized Controlled Trial
Brief Title: Timing of Complete Revascularization in Patients With ST-segment Elevation Myocardial Infarction And Multivessel Disease
Acronym: TERMINAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: Beijing Chao Yang Hospital (Other); Beijing Luhe Hospital (Other)
Responsible Party: Principal Investigator, Xiaotong Hou, Clinical Professor, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-20
Record Dates: First submitted 2021-12-30; First posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: ST-elevation Myocardial Infarction; Multivessel Coronary Disease
Keywords: Acute ST segment elevation myocardial infarction; Multi vessel lesions; Complete revascularization; Non infarct related arteries; Major cardiovascular adverse events
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediately CR group (Experimental): Immediately open non-IRA after successful emergency PCI of IRA in STEMI patients with MVD
  Interventions: Procedure: Immediately CR
- Staged (within 45 days) CR group (Active Comparator): Strategy of opening non-IRA by stages after emergency PCI of IRA in STEMI patients with MVD
  Interventions: Procedure: Staged (within 45 days) CR

INTERVENTIONS:
Procedure: Immediately CR — Immediately opening non-IRA after emergency opening IRA in STEMI patients with MVD
  Arms: Immediately CR group
Procedure: Staged (within 45 days) CR — Staged opening non-IRA after emergency opening IRA in STEMI patients with MVD
  Arms: Staged (within 45 days) CR group

SUMMARY:
At present, the two treatment strategies of opening non infarct related arteries (non IRA) simultaneously or by stages after emergency percutaneous coronary intervention (PCI) in patients with acute ST segment elevation myocardial infarction (STEMI) complicated with multi vessel disease (MVD) are still controversial. In our previous retrospective analysis, there was no significant difference between complete revascularization (CR) and staged CR at Anzhen Hospital in the cases of cardiac death, reinfarction, stroke, proportion of revascularization and hospitalization rate of heart failure.

DETAILED DESCRIPTION:
The literature reports on the benefits of two CR strategies of opening non IRA simultaneously or by stages after IRA treatment in STEMI patients are inconsistent. This study intends to enroll 426 cases and divide into two groups to verify whether the occurrence of major cardiovascular adverse events (all-cause death, nonfatal myocardial infarction, ischemia driven revascularization and heart failure) in one year in immediately open non-IRA after successful emergency PCI of infarct related arteries in STEMI patients with MVD group is not inferior to staged (within 45 days) CR group. It can accumulate more evidence-based medical basis for the selection of better treatment schemes, so as to formulate optimized treatment schemes for clinic. To study when to open meaningful non IRA in acute STEMI complicated with MVD is of great guiding significance for CR after acute myocardial infarction. At the same time, it has important social significance and economic value for delaying or preventing cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

1. Onset of the spontaneous acute STEMI (24 hours).
2. The anatomical structure of coronary artery is suitable for complete revascularization by PCI.
3. It is suitable for PCI through radial artery or femoral artery.
4. Be able to fully identify Infarct-related artery（IRA）.
5. In addition to IRA, in the vessels of lumen diameter is 2.25mm or more, but less than 4.5mm. there is at least one non IRA's stenosis more than 70% observed in both planes, or 50% ~ 69% stenosis and fractional flow reserve (FFR) or Quantitative Flow Ratio (QFR) measured value is 0.80 or less.
6. After IRA revascularization the thrombolysis in myocardial infarction (TIMI) blood flow is in grade 3.
7. The hemodynamics of patients after IRA revascularization is stable, that is, systolic blood pressure ≥ 90mmHg, or blood pressure ≥ 90mmHg after catecholamines, and there is no clinical manifestation of hypoperfusion.
8. Patient who has signed informed consent

Exclusion Criteria:

1. Cardiogenic shock which means a group of clinical syndromes leading to cardiac dysfunction caused by various reasons, which meet the following criteria: A: continuous hypotension, systolic blood pressure < 90mmHg or mean arterial pressure decreased from baseline ≥ 30mmhg, more than 30min; B: cardiac index < 1.8l/min/m2, pulmonary congestion or elevated left ventricular filling pressure; c: Signs of organ perfusion damage (at least one): changes in mental state, wet and cold skin, oliguria, and increased serum lactic acid level.
2. The duration of cardiopulmonary resuscitation is more than 10 minutes.
3. Emergency coronary artery bypass grafting (CABG) is needed.
4. Previous coronary-artery bypass grafting surgery.
5. Hybrid revascularization is planned.
6. Coronary dissection.
7. Stent thrombosis.
8. In stent restenosis, definition: A: target vessel diameter stenosis ≥ 50% at follow-up. b: The lumen loss at follow-up was larger than 50% of the net lumen gain after operation. c: The lumen diameter at follow-up and the minimum diameter loss measured immediately at stenting were 0.72 mm or more.
9. Acute myocardial infarction complicated with severe mechanical complications, defined as acute severe mitral regurgitation, ventricular septal perforation and cardiac free wall rupture / pericardial tamponade.
10. Severe renal failure (EGFR < 30ml / min) or dialysis treatment is required.
11. Chronic total occlusion of main coronary artery.
12. Complex bifurcation lesions requiring dual stent treatment.
13. Stenosis of Left main coronary artery≥ 50% or stenosis of left anterior descending coronary artery and circumflex coronary artery ≥ 70%.
14. Coronary, cerebrovascular or peripheral revascularization is planned.
15. Cardiac surgery or other surgical treatment is planned.
16. Contraindications to double antibody therapy [aspirin and P2Y12 inhibitor (clopidogrel or ticagrelor) for 3 months.
17. pregnant woman.
18. Patient who has participated in other clinical trials.
19. Life expectancy < 1 year.
20. Patient who is not suitable for inclusion in the study according to the operator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Event | 1 year
  Including All-cause death, Ischemia driven revascularization, Nonfatal myocardial infarction and Heart failure

SECONDARY OUTCOMES:
All-cause death | 1 year
  All reasons of death
Ischemia driven revascularization | 1 year
  Myocardial ischemia needs to revascularize
Nonfatal myocardial infarction | 1 year
  A kind of Myocardial infarction which does not lead to death
Heart failure | 1 year
  Deterioration of heart function or acute heart failure
Cardiovascular related death | 1 year
  Died of cardiovascular diseases
Stent thrombosis | 1 year
  Thrombosis in stent
Dialysis or acute renal insufficiency | 1 year
  Dialysis or acute renal insufficiency occurred after operation
Bleeding events | 1 year
  Bleeding occurred after oral administration of dual antiplatelet drugs

CONTACTS AND LOCATIONS:
Overall Officials: Hou, Study Director — Beijing Anzhen Hospital
Locations (1):
- Center for Cardiac Intensive Care, Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ibanez B, Roque D, Price S. The year in cardiovascular medicine 2020: acute coronary syndromes and intensive cardiac care. Eur Heart J. 2021 Mar 1;42(9):884-895. doi: 10.1093/eurheartj/ehaa1090. No abstract available. PMID 33388774
- [Background] Park DW, Clare RM, Schulte PJ, Pieper KS, Shaw LK, Califf RM, Ohman EM, Van de Werf F, Hirji S, Harrington RA, Armstrong PW, Granger CB, Jeong MH, Patel MR. Extent, location, and clinical significance of non-infarct-related coronary artery disease among patients with ST-elevation myocardial infarction. JAMA. 2014 Nov 19;312(19):2019-27. doi: 10.1001/jama.2014.15095. PMID 25399277
- [Background] Sorajja P, Gersh BJ, Cox DA, McLaughlin MG, Zimetbaum P, Costantini C, Stuckey T, Tcheng JE, Mehran R, Lansky AJ, Grines CL, Stone GW. Impact of multivessel disease on reperfusion success and clinical outcomes in patients undergoing primary percutaneous coronary intervention for acute myocardial infarction. Eur Heart J. 2007 Jul;28(14):1709-16. doi: 10.1093/eurheartj/ehm184. Epub 2007 Jun 7. PMID 17556348
- [Background] Politi L, Sgura F, Rossi R, Monopoli D, Guerri E, Leuzzi C, Bursi F, Sangiorgi GM, Modena MG. A randomised trial of target-vessel versus multi-vessel revascularisation in ST-elevation myocardial infarction: major adverse cardiac events during long-term follow-up. Heart. 2010 May;96(9):662-7. doi: 10.1136/hrt.2009.177162. Epub 2009 Sep 23. PMID 19778920
- [Background] Hannan EL, Samadashvili Z, Walford G, Holmes DR Jr, Jacobs AK, Stamato NJ, Venditti FJ, Sharma S, King SB 3rd. Culprit vessel percutaneous coronary intervention versus multivessel and staged percutaneous coronary intervention for ST-segment elevation myocardial infarction patients with multivessel disease. JACC Cardiovasc Interv. 2010 Jan;3(1):22-31. doi: 10.1016/j.jcin.2009.10.017. PMID 20129564
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Background] Montone RA, Niccoli G, Crea F, Jang IK. Management of non-culprit coronary plaques in patients with acute coronary syndrome. Eur Heart J. 2020 Oct 1;41(37):3579-3586. doi: 10.1093/eurheartj/ehaa481. PMID 32676644
- [Background] Wald DS, Morris JK, Wald NJ, Chase AJ, Edwards RJ, Hughes LO, Berry C, Oldroyd KG; PRAMI Investigators. Randomized trial of preventive angioplasty in myocardial infarction. N Engl J Med. 2013 Sep 19;369(12):1115-23. doi: 10.1056/NEJMoa1305520. Epub 2013 Sep 1. PMID 23991625
- [Background] Gershlick AH, Khan JN, Kelly DJ, Greenwood JP, Sasikaran T, Curzen N, Blackman DJ, Dalby M, Fairbrother KL, Banya W, Wang D, Flather M, Hetherington SL, Kelion AD, Talwar S, Gunning M, Hall R, Swanton H, McCann GP. Randomized trial of complete versus lesion-only revascularization in patients undergoing primary percutaneous coronary intervention for STEMI and multivessel disease: the CvLPRIT trial. J Am Coll Cardiol. 2015 Mar 17;65(10):963-72. doi: 10.1016/j.jacc.2014.12.038. PMID 25766941
- [Background] Engstrom T, Kelbaek H, Helqvist S, Hofsten DE, Klovgaard L, Holmvang L, Jorgensen E, Pedersen F, Saunamaki K, Clemmensen P, De Backer O, Ravkilde J, Tilsted HH, Villadsen AB, Aaroe J, Jensen SE, Raungaard B, Kober L; DANAMI-3-PRIMULTI Investigators. Complete revascularisation versus treatment of the culprit lesion only in patients with ST-segment elevation myocardial infarction and multivessel disease (DANAMI-3-PRIMULTI): an open-label, randomised controlled trial. Lancet. 2015 Aug 15;386(9994):665-71. doi: 10.1016/s0140-6736(15)60648-1. PMID 26347918
- [Background] Smits PC, Abdel-Wahab M, Neumann FJ, Boxma-de Klerk BM, Lunde K, Schotborgh CE, Piroth Z, Horak D, Wlodarczak A, Ong PJ, Hambrecht R, Angeras O, Richardt G, Omerovic E; Compare-Acute Investigators. Fractional Flow Reserve-Guided Multivessel Angioplasty in Myocardial Infarction. N Engl J Med. 2017 Mar 30;376(13):1234-1244. doi: 10.1056/NEJMoa1701067. Epub 2017 Mar 18. PMID 28317428
- [Background] Kornowski R, Mehran R, Dangas G, Nikolsky E, Assali A, Claessen BE, Gersh BJ, Wong SC, Witzenbichler B, Guagliumi G, Dudek D, Fahy M, Lansky AJ, Stone GW; HORIZONS-AMI Trial Investigators. Prognostic impact of staged versus "one-time" multivessel percutaneous intervention in acute myocardial infarction: analysis from the HORIZONS-AMI (harmonizing outcomes with revascularization and stents in acute myocardial infarction) trial. J Am Coll Cardiol. 2011 Aug 9;58(7):704-11. doi: 10.1016/j.jacc.2011.02.071. PMID 21816305
- [Background] Manari A, Varani E, Guastaroba P, Menozzi M, Valgimigli M, Menozzi A, Magnavacchi P, Franco N, Marzocchi A, Casella G. Long-term outcome in patients with ST segment elevation myocardial infarction and multivessel disease treated with culprit-only, immediate, or staged multivessel percutaneous revascularization strategies: Insights from the REAL registry. Catheter Cardiovasc Interv. 2014 Nov 15;84(6):912-22. doi: 10.1002/ccd.25374. Epub 2014 Feb 1. PMID 24403174